CLINICAL TRIAL: NCT03561142
Title: Organ Preservation in Locally Advanced Rectal Cancer by Radiochemotherapy Followed by Consolidation Chemotherapy. A Prospective Phase II Pilot Trial of the German Rectal Cancer Study Group
Brief Title: Organ Preservation in Locally Advanced Rectal Cancer by Radiochemotherapy Followed by Consolidation Chemotherapy.
Acronym: CAO/ARO/AIO-16
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAOAROAIO16
Record Dates: First submitted 2018-04-19; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Rectal Cancer; Rectal Neoplasms; Rectal Cancer Stage II; Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients will undergo different treatments based on response achieved after radiochemotherapy.
  1. Clinical Complete Response: Omission of surgery and follow-up
  2. Near clinical complete response: Reevaluation in three months
  3. Poor / no response: Surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiochemotherapy -> chemotherapy. (Experimental): Radiochemotherapy followed by consolidation chemotherapy. Deep regional hyperthermia can additionally be performed at the centers in Tübingen and Erlangen.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy; Other: Deep regional hyperthermia

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy: 28 x 1.8 Gy (total: 50.4 Gy), 5 fractions per week on day 1- 38
Drug: Chemotherapy — chemoradiotherapy is started according to the following schedule: 5-FU: 250 mg/sqm per day, iv, on day 1-14, day 22-35; Oxaliplatin: 50 mg/sqm, day 1, 8, 22, and 29. After a break of two and a half weeks, patients receive three chemotherapy cycles, starting on day 57, 71 and 85, consisting of: Folinic acid: 400 mg/sqm, 2h-iv; Oxaliplatin: 100 mg/sqm, 2h-iv; 5-FU: 2400 mg/sqm, 46h-iv
  Other Names: all brands of the used drugs are allowed
Other: Deep regional hyperthermia — Deep regional hyperthermia to the pelvis, total time 90 min, target temperature 41-42°C. Twice weekly, up to a total of 10 sessions within d1 and d38.
  Deep regional hyperthermia is offered at the centers in Tübingen and Erlangen.

SUMMARY:
There is a growing body of evidence that surgery and associated morbidities can be omitted without compromising oncological safety in selected patients who have achieved a clinical complete response after radiochemotherapy. However with standard neoadjuvant treatment regimens the pathological complete response rate lies in the range between 10%-20%, the number of patients qualifying for non-operative management is even lower since the sensitivity of currently available diagnostic measures for predicting the pathological complete response hardly surpasses 50%-60%.The hereby proposed phase II trial CAO/ARO/AIO-16 aims at finding novel and innovative aspects of rectal cancer treatment. According to recently published data the radiochemotherapy regime in the present study with consolidating chemotherapy and delayed assessment of response has the potential to achieve pathological complete rates of approximately 40%. A standardized re-evaluation after consolidating chemotherapy will select patients who are candidates for organ-preservation. These patients will not undergo radical surgery and will instead be follow-up closely for tumor regrowth.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with histologically confirmed diagnosis of rectal cancer localized 0 - 12 cm from the anocutaneous line as measured by rigid rectoscopy (i.e. lower and middle third of the rectum)
* Any MRI staged cT3 tumor or any cT1 cN+ or cT2 cN+ with nodal staging according to "SOP MRI"
* Staging requirements: High-resolution, thin-sliced (i.e. 3mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* Cross-sectional imaging of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit.
* WHO/ECOG Performance Status ≤ 1
* Adequate hematological, hepatic, renal and metabolic function parameters
* Informed consent of the patient

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm from the anocutaneous line as measured by rigid rectoscopy
* cT4 tumors
* Positive lateral pelvic lymph nodes
* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* Preexisting fecal incontinence for solid stool
* Preexisting peripheral sensory neuropathy with functional impairment
* Preexisting myelosuppression reflected by a neutrophil count < 2.000/mm^3 and/or platelets < 100.000/mm^3
* Severe impairment of kidney function with a Creatinin Clearance < 30 ml/min)
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception according to the "Clinical trial fertility group"
* On-treatment participation in an interventional clinical study in the period 30 days prior to inclusion
* Previous or current drug abuse
* Other concomitant antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder, severe liver function disorders
* WHO/ECOG Performance Status > 1
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment.
* Chronic diarrhea (> grade 1 according NCI CTCAE) Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1), if the patient is continuously disease-free
* Known allergic reactions on study medication
* Known dihydropyrimidine dehydrogenase deficiency
* Medication inhibitors of the dihydropyrimidine dehydrogenase, such as Brivudin, Sorivudin and its analogues.
* Pernicious anemia or other anemias caused by Vitamin B-12 deficiency.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).
* Additionally for hyperthermia cardiac pacemakers and metal implants in the proximity of the pelvis constitute a criterion for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2020-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response rate | Day 106 after the start of treatment
  Response to treatment is assessed on day 106 after the start of radiochemotherapy.
  A clinical complete response is defined by standardized findings in rectoscopy, MRI and digital rectal examination

SECONDARY OUTCOMES:
Local regrowth rate | 4 years
Safety of the treatment (toxicity assessment according to NCI CTCAE Version 4.0) | 4 years
Fecal incontinence according to Wexner-Vaizey Score | 4 years
  Possible scores range from 0 (perfect continence) to 24 (complete incontinence)
Quality of life according to EORTC Quality of Life questionnaire - C30 | 4 years
Quality of life according to EORTC Quality of Life questionnaire - CR29 | 4 years
Frequency of Low anterior resection syndrome (LARS-scale) | 4 years
Surgical morbidity in patients undergoing surgery | up to 30 days after surgery
Surgical complications in patients undergoing surgery | up to 30 days after surgery
Pathological staging, tumor downstaging (assessed by ypTNM findings in relation to initial cTNM staging), tumor regression grading according to Dworak in patients undergoing surgery | Day 123 after the start of treatment
R0 resection rate, rate of circumferential resection margin negativity (> 1mm) in patients undergoing surgery | Day 123 after the start of treatment
Rate of sphincter-sparing surgery in patients undergoing surgery | Day 123 after the start of treatment
Relapse-free survival (local / distant / overall) | 4 years
Overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Gani, Dr., Principal Investigator — University Hospital Tübingen
Locations (4):
- Germany (4):
  - University Hospital Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Tübingen, Tübingen
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gani C, Bonomo P, Zwirner K, Schroeder C, Menegakis A, Rodel C, Zips D. Organ preservation in rectal cancer - Challenges and future strategies. Clin Transl Radiat Oncol. 2017 Mar 23;3:9-15. doi: 10.1016/j.ctro.2017.02.002. eCollection 2017 Apr. PMID 29658007
- [Background] Schroeder C, Gani C, Lamprecht U, von Weyhern CH, Weinmann M, Bamberg M, Berger B. Pathological complete response and sphincter-sparing surgery after neoadjuvant radiochemotherapy with regional hyperthermia for locally advanced rectal cancer compared with radiochemotherapy alone. Int J Hyperthermia. 2012;28(8):707-14. doi: 10.3109/02656736.2012.722263. Epub 2012 Sep 24. PMID 23006132
- [Background] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Derived] Gani C, Fokas E, Polat B, Ott OJ, Diefenhardt M, Konigsrainer A, Boke S, Kirschniak A, Bachmann R, Wichmann D, Bitzer M, Clasen S, Grosse U, Hoffmann R, Gotz M, Hofheinz RD, Germer E, Germer CT, Fietkau R, Martus P, Zips D, Rodel C. Organ preservation after total neoadjuvant therapy for locally advanced rectal cancer (CAO/ARO/AIO-16): an open-label, multicentre, single-arm, phase 2 trial. Lancet Gastroenterol Hepatol. 2025 Jun;10(6):562-572. doi: 10.1016/S2468-1253(25)00049-4. PMID 40347958